CLINICAL TRIAL: NCT05820828
Title: Does Venous Cannulation Method Affect Air Embolic Load to the Patient During Extracorporeal Circulation?
Brief Title: Comparing Air Embolic Load in Two Venous Cannulation Methods, 40 Patients Undergoing Elective Valve Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petronella Torild (Other)
Responsible Party: Sponsor-Investigator, Petronella Torild, Perfusionist aspirant, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-00204-01
Record Dates: First submitted 2023-03-16; First posted 2023-04-20 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Extracorporeal Circulation; Complications; Air Embolism
MeSH Terms: conditions — Embolism, Air

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patient will during extracorporeal circulation be monitored and held in the range of > 300 mL in the venous reservoir. Patient will recieve fluid if needed to maintain correct level (crystalloids, colloids or erytrocytes depending on patients clinical status).
- Interventional group (Experimental): Patient will during extracorporeal circulation be monitored and held in the range of 200 - 300 mL in the venous reservoir. To maintain correct level of volume, any excessive fluid will be drained into a sterile infusion bag during extracorporeal circulation. After the surgery, the patient will recieve the volume to ensure correct volume status.
  Interventions: Diagnostic Test: Volume control

INTERVENTIONS:
Diagnostic Test: Volume control — Volume control in venous reservoir during extracorporeal circulation.
  Arms: Interventional group

SUMMARY:
The goal of this single center prospective controlled observational and interventional trial is to investigate and compare origin of air emboli when different venous cannulation methods is used in patients undergoing cardiac surgery with extracorporeal circulation.

40 consecutive elective patients will be included in two groups, depending on the procedure requiring bicaval or cavoatrial cannulation. After assorted into respective group, patients will be block randomized (five groups consisting of eight patients each) to either intervention group (low venous reservoir volume, 200-300 mL) or control group (venous reservoir volume > 300 mL).

Primary endpoint is to investigate if the amount of air emboli passing through the oxygenator to the arterial line differs between bicaval and cavoatrial venous cannulation during extracorporeal circulation. Secondary endpoints are the relative difference in amount air emboli between the groups, if there is any correlation between the amount of air in venous line and the amount of air passing through the oxygenator to the arterial line during extracorporeal circulation, and if difference is seen on the amount of air passing through the oxygenator depending on the level of volume in the venous reservoir.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years
* Elective bicaval cannulation (mitral valve repair/replacement (MVR) or MVR + coronary artery bypass grafting (CABG))
* Elective cavoatrial cannulation (aortic valve repair/replacement (AVR) or AVR + CABG
* Planned normothermia (35-37˚C)

Exclusion Criteria:

* Acute heart surgery
* Adult Congenital Heart Disease (ACHD) surgery
* Endocarditis
* Reoperation (primary procedure > 2 years ago)
* Perioperative iatrogenic adverse events (major bleeding, aortic dissection, other severe complications)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Difference in count (number) of air emboli passing through the oxygenator to the arterial line between bicaval and cavoatrial venous cannulation. | 1 day (During extracorporeal circulation)
  Bubble counter measurements
Difference in volume (nano liter) of air emboli passing through the oxygenator to the arterial line between bicaval and cavoatrial venous cannulation. | 1 day (During extracorporeal circulation)
  Bubble counter measurements

SECONDARY OUTCOMES:
Difference in the amount of air emboli in venous tubing between bicaval and cavoatrial cannulation. | 1 day (During extracorporeal circulation)
  Bubble counter measurements
Correlation between the amount of air in venous line and the amount of air passing through the oxygenator to the arterial line during extracorporeal circulation. | 1 day (During extracorporeal circulation)
  Bubble counter measurements
Difference in amount of air passing through the oxygenator depending on the volume in the venous reservoir (200-300 mL versus > 300 mL). | 1 day (During extracorporeal circulation)
  Bubble counter measurements

CONTACTS AND LOCATIONS:
Overall Officials: Tor Damen, PhD, Principal Investigator — Dep of Anesthesiology and Intensive Care Medicine, Sahlgrenska University Hospital
Locations (1):
- Department of Cardiothoracic Surgery, Perfusion. Sahlgrenska University Hospital., Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Torild P, Corderfeldt Keiller A, Damen T. Does the venous cannulation method affect gaseous embolic load to the patient during extracorporeal circulation? Perfusion. 2026 Jan;41(1):102-109. doi: 10.1177/02676591251344859. Epub 2025 May 20. PMID 40393695